CLINICAL TRIAL: NCT05138406
Title: The Effect of Graded Motor Imagery Training on Pain, Functional Performance, Motor Imagery Skill, and Kinesiophobia After Total Knee Arthroplasty.
Brief Title: Graded Motor Imagery and Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burcu Talu, Associate professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/173
Record Dates: First submitted 2021-10-28; First posted 2021-12-01 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Total Knee Arthroplasty
Keywords: Graded Motor Imagery; Pain; Rehabilitation; Total knee arthroplasty
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graded Motor Imagery (Experimental): Individuals will receive standard rehabilitation and graded motor imagery treatment.
  Interventions: Other: Graded Motor Imagery; Other: Standard Rehabilitation
- Standard Rehabilitation Group (Active Comparator): Standard rehabilitation will be applied.
  Interventions: Other: Standard Rehabilitation

INTERVENTIONS:
Other: Graded Motor Imagery — The graded motor imaging program will be set to 2 weeks each component. Participants will receive lateralization for the first 2 weeks, motor imagery for 2 weeks, and mirror therapy for 2 weeks. At the same time, standard rehabilitation will be applied for 6 weeks. Treatments will begin 24-48 hours after surgery. Treatments will be applied under the control of a physiotherapist 3 days a week and as home exercise 3 days a week.
  Arms: Graded Motor Imagery
Other: Standard Rehabilitation — Standard rehabilitation consisting of cold therapy, stretching and strengthening exercises will be applied. Treatment will be applied under the control of a physiotherapist 3 days a week and as home exercise 3 days a week.

SUMMARY:
This study was planned to investigate the long-term effectiveness of the early application of graded motor imagery therapy on pain parameters, functional performance, motor imagery skill, and kinesiophobia in individuals who underwent total knee arthroplasty surgery after knee osteoarthritis.

DETAILED DESCRIPTION:
Participants aged 45-80 who are scheduled for total knee arthroplasty surgery after knee osteoarthritis will be included. Participants will be selected from the relevant population using a nonprobability random sampling method. Participants who agree to participate in the study and meet the inclusion criteria will be assigned to one of the groups (conventional rehabilitation-only or conventional rehabilitation with graded motor imagery) using the closed envelope method. Evaluations will be made one day before surgery, 6 weeks and 6 months after surgery for each group. Pain Visual Analog Scale; pressure pain threshold algometer; central sensitization Central Sensitization Inventory; the joint range of motion goniometer; muscle strength handheld dynamometer; kinesiophobia Tampa Kinesiophobia Scale; functional mobility and mental stopwatch Timed get up and go test; choice task Recognise™ application; motor imagery skill Movement Imagery Questionnaire-3; functional assessment Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC); The catastrophic degree of pain is planned to be evaluated with the Pain Catastrophizing Scale.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee osteoarthritis and being on the waiting list to receive unilateral total knee arthroplasty
* Approved by the orthopedist for early physiotherapy treatment after total knee arthroplasty

Exclusion Criteria:

* - Individuals undergoing revision total knee arthroplasty or undergoing bilateral total knee arthroplasty,
* Contralateral knee osteoarthritis (defined by activity greater than 4/10 pain)
* Having undergone any physical therapy intervention or other surgery in the last 6 months
* Any neurological, cardiac, pulmonary or psychiatric disease (eg, uncontrolled diabetes mellitus, neoplasms, uncontrolled blood pressure, neurological conditions) before or after surgery;
* Fracture, infection in the acute postoperative phase or presence of fever
* Cognitive impairments that alter the probability of correct understanding of the motor imagery program
* Body mass index > 35 kg / m2
* Difficulties with understanding or communication
* Insufficient knowledge of Turkish to follow the study instructions.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline
  Pain at rest and during activity will be evaluated with the help of the Visual Analogue Scale (VAS). The VAS is a 10 cm scale that rates 0 points as "no pain" and 10 points as "worst pain imaginable".
Pain intensity | 6 weeks after surgery
  Pain at rest and during activity will be evaluated with the help of the Visual Analogue Scale (VAS). The VAS is a 10 cm scale that rates 0 points as "no pain" and 10 points as "worst pain imaginable".
Pain intensity | 6 months after surgery
  Pain at rest and during activity will be evaluated with the help of the Visual Analogue Scale (VAS). The VAS is a 10 cm scale that rates 0 points as "no pain" and 10 points as "worst pain imaginable".
WOMAC | Baseline
  Functional status will be assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). It consists of three subgroups as pain (5 items), stiffness (2 items) and physical function (17 items) and a total of 24 items. Each item has an evaluation score of 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe.
WOMAC | 6 weeks after surgery
  Functional status will be assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). It consists of three subgroups as pain (5 items), stiffness (2 items) and physical function (17 items) and a total of 24 items. Each item has an evaluation score of 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe.
WOMAC | 6 months after surgery
  Functional status will be assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). It consists of three subgroups as pain (5 items), stiffness (2 items) and physical function (17 items) and a total of 24 items. Each item has an evaluation score of 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe.

SECONDARY OUTCOMES:
Pressure pain threshold | Baseline
  A pressure algometer (digital algometer) will be used. It will be evaluated at four test sites at the knee (medial and lateral edge of the patella, lateral and medial femoral condyles) and one distal painless zone at the wrist extensors (5 cm distal to the lateral epicondyle).
  It will be pressed with increasing pressure and the individual will be asked to say "yes" as soon as the participant feels pain or discomfort. Three attempts will be made at each point with a 30-second rest and the averages recorded.
Pressure pain threshold | 6 weeks after surgery
  A pressure algometer (digital algometer) will be used. It will be evaluated at four test sites at the knee (medial and lateral edge of the patella, lateral and medial femoral condyles) and one distal painless zone at the wrist extensors (5 cm distal to the lateral epicondyle).
  It will be pressed with increasing pressure and the individual will be asked to say "yes" as soon as the participant feels pain or discomfort. Three attempts will be made at each point with a 30-second rest and the averages recorded.
Pressure pain threshold | 6 months after surgery
  A pressure algometer (digital algometer) will be used. It will be evaluated at four test sites at the knee (medial and lateral edge of the patella, lateral and medial femoral condyles) and one distal painless zone at the wrist extensors (5 cm distal to the lateral epicondyle).
  It will be pressed with increasing pressure and the individual will be asked to say "yes" as soon as the participant feels pain or discomfort. Three attempts will be made at each point with a 30-second rest and the averages recorded.
Central sensitization | Baseline
  It will be evaluated with the Central Sensitization Inventory. It consists of 2 parts, part A, which evaluates the symptoms thought to be associated with central sensitization syndromes, and part B, which quickly questions whether the patient has received a specific diagnosis before. In part A, there are 25 items that question the frequency of symptoms seen in central sensitization syndromes and are scored between 0-100 points. Each symptom is defined as "never" (0 points) if the patient never experiences that symptom, "rarely" (1 point) if rarely, "sometimes" if sometimes (2 points), "frequently" (3 points) if often It is recorded as "always" (4 points). As the patient's central sensitization inventory score increases, it is thought that he has more symptoms related to central sensitization. In part B, it is questioned whether the patient has ever been diagnosed with any of the diseases included in the central sensitization syndromes by any physician.
Central sensitization | 6 weeks after surgery
  It will be evaluated with the Central Sensitization Inventory. It consists of 2 parts, part A, which evaluates the symptoms thought to be associated with central sensitization syndromes, and part B, which quickly questions whether the patient has received a specific diagnosis before. In part A, there are 25 items that question the frequency of symptoms seen in central sensitization syndromes and are scored between 0-100 points. Each symptom is defined as "never" (0 points) if the patient never experiences that symptom, "rarely" (1 point) if rarely, "sometimes" if sometimes (2 points), "frequently" (3 points) if often It is recorded as "always" (4 points). As the patient's central sensitization inventory score increases, it is thought that he has more symptoms related to central sensitization. In part B, it is questioned whether the patient has ever been diagnosed with any of the diseases included in the central sensitization syndromes by any physician.
Central sensitization | 6 months after surgery
  It will be evaluated with the Central Sensitization Inventory. It consists of 2 parts, part A, which evaluates the symptoms thought to be associated with central sensitization syndromes, and part B, which quickly questions whether the patient has received a specific diagnosis before. In part A, there are 25 items that question the frequency of symptoms seen in central sensitization syndromes and are scored between 0-100 points. Each symptom is defined as "never" (0 points) if the patient never experiences that symptom, "rarely" (1 point) if rarely, "sometimes" if sometimes (2 points), "frequently" (3 points) if often It is recorded as "always" (4 points). As the patient's central sensitization inventory score increases, it is thought that he has more symptoms related to central sensitization. In part B, it is questioned whether the patient has ever been diagnosed with any of the diseases included in the central sensitization syndromes by any physician.
Joint Range of Motion | Baseline
  Active knee flexion and extension angle will be evaluated.
Joint Range of Motion | 6 weeks after surgery
  Active knee flexion and extension angle will be evaluated.
Joint Range of Motion | 6 months after surgery
  Active knee flexion and extension angle will be evaluated.
Quadriceps muscle strength | Baseline
  It will be measured during maximum voluntary isometric contraction using a hand-held muscle tester. After a warm-up test attempt, participants will be asked to extend their knees with maximum force against the device for five seconds. Two trials separated by a rest period of 120 seconds will be performed and averaged.
Quadriceps muscle strength | 6 weeks after surgery
  It will be measured during maximum voluntary isometric contraction using a hand-held muscle tester. After a warm-up test attempt, participants will be asked to extend their knees with maximum force against the device for five seconds. Two trials separated by a rest period of 120 seconds will be performed and averaged.
Quadriceps muscle strength | 6 months after surgery
  It will be measured during maximum voluntary isometric contraction using a hand-held muscle tester. After a warm-up test attempt, participants will be asked to extend their knees with maximum force against the device for five seconds. Two trials separated by a rest period of 120 seconds will be performed and averaged.
Kinesiophobia | Baseline
  The Tampa Kinesiophobia Scale will be used. A 4-point Likert score (1=I totally disagree, 2=Agree, 3=Disagree, 4=Totally agree) is used for each question in the scale. As a result of the survey, the person gets a total score between 17-68. A high score on the scale indicates a high level of kinesiophobia.
Kinesiophobia | 6 weeks after surgery
  The Tampa Kinesiophobia Scale will be used. A 4-point Likert score (1=I totally disagree, 2=Agree, 3=Disagree, 4=Totally agree) is used for each question in the scale. As a result of the survey, the person gets a total score between 17-68. A high score on the scale indicates a high level of kinesiophobia.
Kinesiophobia | 6 months after surgery
  The Tampa Kinesiophobia Scale will be used. A 4-point Likert score (1=I totally disagree, 2=Agree, 3=Disagree, 4=Totally agree) is used for each question in the scale. As a result of the survey, the person gets a total score between 17-68. A high score on the scale indicates a high level of kinesiophobia.
Functional mobility | Baseline
  The Timed Up and Go test will be used. While the patient is sitting in a chair; will be asked to get up from the chair, walk 3 meters as fast as possible, turn around and sit back in the chair. The time elapsed while the patient performs the test will be recorded.
Functional mobility | 6 weeks after surgery
  The Timed Up and Go test will be used. While the patient is sitting in a chair; will be asked to get up from the chair, walk 3 meters as fast as possible, turn around and sit back in the chair. The time elapsed while the patient performs the test will be recorded.
Functional mobility | 6 months after surgery
  The Timed Up and Go test will be used. While the patient is sitting in a chair; will be asked to get up from the chair, walk 3 meters as fast as possible, turn around and sit back in the chair. The time elapsed while the patient performs the test will be recorded.
Mental chronometry delta time | Baseline
  Timed Get Up and Go test will be used. It compares the time between the actual movement time and the imagined similar task time. At the end of the tests, mental chronometer measurements are calculated in terms of delta time with the formula '(real movement-imagined movement)/[(real movement+imagined movement)/2]x100'.
Mental chronometry delta time | 6 weeks after surgery
  Timed Get Up and Go test will be used. It compares the time between the actual movement time and the imagined similar task time. At the end of the tests, mental chronometer measurements are calculated in terms of delta time with the formula '(real movement-imagined movement)/[(real movement+imagined movement)/2]x100'.
Mental chronometry delta time | 6 months after surgery
  Timed Get Up and Go test will be used. It compares the time between the actual movement time and the imagined similar task time. At the end of the tests, mental chronometer measurements are calculated in terms of delta time with the formula '(real movement-imagined movement)/[(real movement+imagined movement)/2]x100'.
Laterality task | Baseline
  Right-left discrimination will be evaluated using the Recognise™ application. The percentage of correct answers and reaction time will be recorded.
Laterality task | 6 weeks after surgery
  Right-left discrimination will be evaluated using the Recognise™ application. The percentage of correct answers and reaction time will be recorded.
Laterality task | 6 months after surgery
  Right-left discrimination will be evaluated using the Recognise™ application. The percentage of correct answers and reaction time will be recorded.
Movement Imagery Questionnaire-3 (MIQ-3) | Baseline
  It is a questionnaire that evaluates the imagery of four movements consisting of knee bending, jumping, arm movement and bending. It consists of three subscales and a total of 12 items evaluating external visual imagery, internal visual imagery, and kinesthetic imagery. Before starting the questionnaire, participants are given definitions of external visual imagery, internal visual imagery, and kinesthetic imagery. Before scoring each movement, the person is asked to perform the movement, then the movement is visualized three times. It is scored on a scale from 1 to 7. 1 point means "very difficult to see/feel", while 7 points means "very easy to see/feel".
Movement Imagery Questionnaire-3 (MIQ-3) | 6 weeks after surgery
  It is a questionnaire that evaluates the imagery of four movements consisting of knee bending, jumping, arm movement and bending. It consists of three subscales and a total of 12 items evaluating external visual imagery, internal visual imagery, and kinesthetic imagery. Before starting the questionnaire, participants are given definitions of external visual imagery, internal visual imagery, and kinesthetic imagery. Before scoring each movement, the person is asked to perform the movement, then the movement is visualized three times. It is scored on a scale from 1 to 7. 1 point means "very difficult to see/feel", while 7 points means "very easy to see/feel".
Movement Imagery Questionnaire-3 (MIQ-3) | 6 months after surgery
  It is a questionnaire that evaluates the imagery of four movements consisting of knee bending, jumping, arm movement and bending. It consists of three subscales and a total of 12 items evaluating external visual imagery, internal visual imagery, and kinesthetic imagery. Before starting the questionnaire, participants are given definitions of external visual imagery, internal visual imagery, and kinesthetic imagery. Before scoring each movement, the person is asked to perform the movement, then the movement is visualized three times. It is scored on a scale from 1 to 7. 1 point means "very difficult to see/feel", while 7 points means "very easy to see/feel".
Pain Catastrophizing Scale | Baseline
  There are 13 states on the scale that describe different feelings and thoughts that may be associated with pain. Participants in each of these situations; 0: None, 1: Mildly, 2: Moderately, 3: Mostly, 4: Always. The total score is between 0-52; It is obtained by summing all 13 items.
Pain Catastrophizing Scale | 6 weeks after surgery
  There are 13 states on the scale that describe different feelings and thoughts that may be associated with pain. Participants in each of these situations; 0: None, 1: Mildly, 2: Moderately, 3: Mostly, 4: Always. The total score is between 0-52; It is obtained by summing all 13 items.
Pain Catastrophizing Scale | 6 months after surgery
  There are 13 states on the scale that describe different feelings and thoughts that may be associated with pain. Participants in each of these situations; 0: None, 1: Mildly, 2: Moderately, 3: Mostly, 4: Always. The total score is between 0-52; It is obtained by summing all 13 items.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu TALU, Principal Investigator — Inonu University
Locations (1):
- Inonu Unıversity, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] La Touche R, Grande-Alonso M, Cuenca-Martinez F, Gonzalez-Ferrero L, Suso-Marti L, Paris-Alemany A. Diminished Kinesthetic and Visual Motor Imagery Ability in Adults With Chronic Low Back Pain. PM R. 2019 Mar;11(3):227-235. doi: 10.1016/j.pmrj.2018.05.025. Epub 2019 Jan 15. PMID 29908933
- [Background] Dilek B, Ayhan C, Yagci G, Yakut Y. Effectiveness of the graded motor imagery to improve hand function in patients with distal radius fracture: A randomized controlled trial. J Hand Ther. 2018 Jan-Mar;31(1):2-9.e1. doi: 10.1016/j.jht.2017.09.004. Epub 2017 Nov 6. PMID 29122370
- [Background] Gurudut P, Jaiswal R. Comparative Effect of Graded Motor Imagery and Progressive Muscle Relaxation on Mobility and Function in Patients with Knee Osteoarthritis: A Pilot Study. Altern Ther Health Med. 2022 Mar;28(3):42-47. PMID 33128533
- [Background] Lee HG, An J, Lee BH. The Effect of Progressive Dynamic Balance Training on Physical Function, The Ability to Balance and Quality of Life Among Elderly Women Who Underwent a Total Knee Arthroplasty: A Double-Blind Randomized Control Trial. Int J Environ Res Public Health. 2021 Mar 3;18(5):2513. doi: 10.3390/ijerph18052513. PMID 33802559